CLINICAL TRIAL: NCT00321347
Title: A Randomized, Placebo Controlled Phase II Study of Parenteral Lidocaine's Ability To Acutely Relieve Opioid Refractory Pain
Brief Title: Intravenous (IV) Lidocaine for Opioid-refractory Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled and clinician no longer at institution.
Sponsor: San Diego Hospice & Palliative Care (Other)
Responsible Party: Principal Investigator, Jay Thomas, Principal Investigator, San Diego Hospice & Palliative Care
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPS-05-002-MI
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Neoplasms; Pain
Keywords: Cancer; Pain; Lidocaine
MeSH Terms: conditions — Neoplasms; Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
Opioid medicines, like morphine, are the main treatment for severe cancer pain. Unfortunately, some patients suffer severe pain despite high doses of opioids. We hypothesize that intravenous lidocaine can quickly and effectively treat this kind of opioid-refractory pain.

DETAILED DESCRIPTION:
Pain is a pervasive symptom among advanced cancer patients. In addition to pain's negative impact, unrelieved pain is linked to depression and precludes patients from dealing with other aspects of life. The World Health Organization 3-step hierarchy for pain management is effective in controlling cancer pain in 70-90% of patients. However, a significant fraction of cancer patients continue to suffer from severe pain despite high dose opioid therapy. This opioid-refractory pain requires adjunctive pain medications. Often multiple adjunctive agents are needed concurrently to optimally control opioid-refractory pain. Unfortunately, patients remain in pain during the time needed to titrate these agents, and some patients don't have this time before their death. Clinically, there exists no widely available, acute intervention to quickly control opioid-refractory pain. Intraspinal delivery of medications, peripheral nerve blocks, and neurolysis help only the subset with well-localized pain syndromes, are invasive, and require subspecialty skills. Sedation quickly relieves pain but robs a patient of the ability to interact. The hypothesis to be tested in this study is that intravenous (IV) lidocaine can acutely palliate opioid-refractory pain. IV lidocaine has been shown to be effective in small trials in non-cancer patients with conditions such as post-herpetic neuralgia and diabetic neuropathy. Additionally, there are case reports of the efficacy of IV lidocaine in cancer patients with opioid-refractory pain. However, there are no randomized, placebo-controlled trials in cancer patients establishing efficacy. Moreover, because of lidocaine's pro-arrhythmic potential and relatively narrow therapeutic window, there is a theoretical risk of harm. As a practical matter of fact, IV lidocaine is not available for the vast majority of cancer patients in the US. To illuminate this situation, a double-blind, randomized, placebo-controlled, study will be conducted to determine the efficacy of IV lidocaine in acutely relieving severe opioid-refractory pain in advanced cancer patients. Secondary end-points include analyses of safety and clinical parameters predictive of lidocaine response. The expected outcome is that lidocaine will acutely, effectively, and safely relieve opioid-refractory pain. This outcome will significantly add to the evidence-based clinical armamentarium available to treat opioid-refractory pain and will significantly improve cancer patients' quality of life.

ELIGIBILITY:
Inclusion Criteria

* Advanced cancer patient (prognosis ≤6 mos)
* Age ≥ 18 years old
* Opioid-refractory pain
* Steady state levels of adjunctive pain medications
* Intravenous access
* Has decision-making capacity
* Hemodynamics: 85<SBP<210 mm Hg & 55<HR<120
* EKG QTc ≤ 440 msec

Exclusion Criteria

* Methadone use
* Myoclonus
* Seizure disorder
* History of ventricular arrhythmia
* Allergy to amide local anesthetics
* Evidence of cardiac ischemia by history or EKG
* Currently receiving a parenteral local anesthetic
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of current pain scores before and after the 30 minute randomized intervention

SECONDARY OUTCOMES:
Preliminary assessment of the safety of intravenous lidocaine
Identify parameters that positively or negatively predict response to lidocaine

CONTACTS AND LOCATIONS:
Overall Officials: Jay R Thomas, MD PhD, Principal Investigator — San Diego Hospice & Palliative Care
Locations (1):
- San Diego Hospice & Palliative Care, San Diego, California, United States